CLINICAL TRIAL: NCT02565940
Title: Study by Metagenomics and Culturomicsapproaches of Bacterial and Viral Flora of Diabetic Foot Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-35
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Diabetic Foot Infection
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic patient with foot infection
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy

SUMMARY:
This work also highlights the presence of an unknown virus double-stranded DNA. In this project we propose 1) incorporating a bank of 150 samples from patients with diabetic foot infection in grades 2-4; 2) to study the microbial flora of a selection of 50 diabetic feet previously untreated with antibiotics for bacterial metagenomics, viral metagenomics and a minimum of 10 per culturomique; 3) to evaluate the use of targeted quantitative PCR on the most frequent new species frequency in the disease and incidentally get a sense of their role in the evolution and prognosis of the disease, including failures of and targeted antibiotic therapy on all 150 samples.

DETAILED DESCRIPTION:
Patients will be included by the infectious and tropical diseases and diabetes services the Nîmes Teaching Hospital which have a large active file and proven expertise internationally in this pathology. The usual agents of infection will be searched by standard bacteriological techniques as part of the microbiological documentation of such cases and will be performed by the microbiology laboratory of CHU Nîmes which will freeze the rest of the sample to -80 ° C the will send it to the Marseille Microbiology Federation for realization of metagenomics-culturomics

ELIGIBILITY:
Inclusion Criteria:

* Patients were taken care by the services(departments) of Diabetology or Infectious diseases of the CHU(TEACHING HOSPITAL) of Nîmes, were hospitalized or were seen in consultation and presenting a wound chronicle of the foot and/or the ankle of Rank 2 - 4 (Classification of the IWGDF) [IWGDF, Lipsky Clin Infect Dis on 2004], inaugural or récidivante.

Exclusion Criteria:

* The patient participates in another study
* The patient is in period of exclusion determined by a previous study
* The patient is under protection(saving) of justice, under guardianship or under guardianship
* The patient refuses to sign the consent
* It turns out impossible to give about the lit(enlightened) information
* The patient is pregnant, parturiente, or she breast-feeds
* The patients having no wound
* The patients diabetics having a wound chronicles of Rank 1 (Classification of the IWGDF) [IWGDF, Lipsky Clin Infect Dis on 2004]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patient with foot infection
Sampling Method: Probability Sample
Enrollment: 150
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
dermal sample | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: desalbres urielle, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Paca, France